CLINICAL TRIAL: NCT03710447
Title: Effects of Concurrent High-Intensity Interval Training and Whole-Body Electromyostimulation on the Cardiometabolic Risk Profile in Obese Individuals at Increased Risk for the Metabolic Syndrome
Brief Title: Effects of Concurrent HIIT and WB-EMS Exercise on the Cardiometabolic Risk Profile in Obese Individuals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COMBI-Study
Record Dates: First submitted 2018-07-01; First posted 2018-10-18 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Overweight and Obesity; Metabolic Syndrome
Keywords: Cardiometabolic Health; Cardiorespiratory Fitness; Muscular Strength; Body Composition; Inflammation; Aerobic Exercise; Resistance Exercise
MeSH Terms: conditions — Overweight; Obesity; Metabolic Syndrome; Inflammation | interventions — galactosylceramide sulfotransferase

STUDY DESIGN:
Intervention Model Description: Parallel Assignment parallel-group, randomized-controlled study
Who Masked: Outcomes Assessor
Masking Description: Outcome Assessors involved in data analysis will not be aware of the arm to which the participants were allocated (single-blinded masking).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HIIT + WB-EMS (Experimental): High-intensity interval training (HIIT) combined with whole-body electromyostimulation (WB-EMS) Sequence of application: HIIT - WB-EMS
  Interventions: Other: HIIT + WB-EMS
- WB-EMS + HIIT (Experimental): Whole-body electromyostimulation (WB-EMS) combined with High-intensity interval training (HIIT) Sequence of application: WB-EMS - HIIT
  Interventions: Other: WB-EMS + HIIT
- HIIT + CST (Experimental): High-intensity interval training (HIIT) combined with conventional low-volume strength training (CST) Sequence of application: HIIT - CST
  Interventions: Other: HIIT + CST
- CST + HIIT (Experimental): Conventional low-volume strength training (CST) combined with high-intensity interval training (HIIT) Sequence of application: CST - HIIT
  Interventions: Other: CST + HIIT

INTERVENTIONS:
Other: HIIT + WB-EMS — 12-week supervised exercise program consisting of ergometer-based high-intensity interval training (HIIT) and whole-body electromyostimulation (WB-EMS).
  HIIT: 5x1 min at 85-95% HRmax divided by low-intensity recovery periods. WB-EMS: Simulanteous stimulation of all major muscle groups with dedicated individual intensity.
  2 exercise sessions per week. Order of application: HIIT - WB-EMS. Additionally, participants receive individualized nutritional counseling.
  Arms: HIIT + WB-EMS
Other: WB-EMS + HIIT — 12-week supervised exercise program consisting of whole-body electromyostimulation (WB-EMS) and ergometer-based high-intensity interval training (HIIT).
  WB-EMS: Simulanteous stimulation of all major muscle groups with dedicated individual intensity.
  HIIT: 5x1 min at 85-95% HRmax divided by low-intensity recovery periods. 2 exercise sessions per week. Order of application: WB-EMS - HIIT. Additionally, participants receive individualized nutritional counseling.
  Arms: WB-EMS + HIIT
Other: HIIT + CST — 12-week supervised exercise program consisting of ergometer-based high-intensity interval training (HIIT) and conventional low-volume strength training(CST).
  HIIT: 5x1 min at 85-95% HRmax divided by low-intensity recovery periods. CST: Conventional 1-set strength training using weight machines to train all major muscle groups with an individual intensity corresponding to 70-80% of one repetition maximum.
  2 exercise sessions per week. Order of application: HIIT - CST. Additionally, participants receive individualized nutritional counseling.
  Arms: HIIT + CST
Other: CST + HIIT — 12-week supervised exercise program consisting of conventional low-volume strength training(CST) and ergometer-based high-intensity interval training (HIIT).
  CST: Conventional 1-set strength training using weight machines to train all major muscle groups with an individual intensity corresponding to 70-80% of one repetition maximum.
  HIIT: 5x1 min at 85-95% HRmax divided by low-intensity recovery periods. 2 exercise sessions per week. Order of application: CST - HIIT. Additionally, participants receive individualized nutritional counseling.
  Arms: CST + HIIT

SUMMARY:
The main purpose of this study is to compare the impact of concurrent high-intensity interval training (HIIT) and whole-body electromyostimulation exercise (WB-EMS) or low-volume conventional strength training (CST) on the cardiometabolic risk profile, overall physical fitness (cardiorespiratory fitness and muscular strength), body composition, inflammatory markers and subjective health outcomes after a 12-week intervention trial in overweight individuals at increased cardiometabolic risk. Furthermore, this study aims to investigate the influence of intra-session exercise order on all outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index >25
* presence of at least 2 cardiometabolic risk factors

Exclusion Criteria:

* Healthy persons or patients under age
* Overweight persons without any additional cardiometabolic risk factors
* Pregnancy, Lactation
* Psychological disorders, epilepsy, sever neurological disorders
* Participation in other exercise- or nutrition studies within the last 6 months
* acute cardiovascular disease
* malignant disease
* Electronic implants (defibrillator, pacemaker)
* Persons in mental hospitals by order of authorities or jurisdiction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-10-15 (Estimated); Primary Completion 2021-10-30 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
Change in Metabolic Syndrome Z-Score (MetS-Z-Score). | 12 weeks
  MetS-Z-Score will be calculated from each individual's measures of waist circumference, mean arterial blood pressure, triglycerides, and HDL-cholesterol, based on equations specific to sex.
Change in overall Physical Fitness Score (PFS) | 12 weeks
  PFS is calculated from VO2max and 1 Repmax values of 5 major muscle Groups.

SECONDARY OUTCOMES:
Change in Body Composition | 12 weeks
  Muscle mass, fat mass and body water will be measured by Bioelectrical Impedance Analysis (BIA)
Change in HOMA-IR | 12 week
  Insulin resistance will be estimated using homeostasis model assessment index (HOMA)
Change Inflammation status | 12 weeks
  Inflammation will be assessed by measuring levels of inflammatory blood markers (CRP, inflammatory cytokines)
Change in Health-related quality of life | 12 weeks
  Health-related quality of life will be assessed by using the standardized and validated EQ-5D-5L Questionnaire
Change in Pain scores | 12 weeks
  Pain scores will be assessed by using the standardized and validated Chronic Pain Grade Questionnaire (CPGQ)
Change in Perceived stress | 12 weeks
  Perceived stress will be assessed by using the standardized and validated Perceived Stress Questionnaire (PSQ)
Change Subjective work ability | 12 weeks
  Subjective work ability will be assessed by using the standardized and validated Work Ability Index Questionnaire (WAI)

CONTACTS AND LOCATIONS:
Overall Officials: Dejan Reljic, Dr., Principal Investigator — University Erlangen Nuremberg Medical School; Yurdaguel Zopf, Prof., Principal Investigator — University Erlangen Nuremberg Medical School
Locations (1):
- Department of Medicine 1, Hector Center for Nutrition, Exercise and Sports, Friedrich-Alexander-University Erlangen-Nuremberg, Erlangen, Germany